CLINICAL TRIAL: NCT05704569
Title: Prediction of Primary Cardiovascular Events Using a Multimarker Approach (Prospective Clinical Study)
Brief Title: Prediction of Primary Cardiovascular Events Using the Multimarker Approach
Status: Completed | Type: Observational
Sponsor: Karaganda Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: CV risk markers
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-01

CONDITIONS: Cardiovascular Diseases; Stroke; Myocardial Infarction; Death; Coronary Artery Disease
Keywords: CVD; biomarkers; prognosis; MI; stroke; CV mortality; CV morbidity
MeSH Terms: conditions — Cardiovascular Diseases; Stroke; Myocardial Infarction; Death; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the outcome group: The composite endpoint included the presence of any of the following events: cardiovascular death, MI, stroke, hospitalization and/or application due to CHD, and transient ischemic attack
  Interventions: Diagnostic Test: measurement of multiple biomarkers
- no-outcome group: individuals who did not experience any events during the observation period
  Interventions: Diagnostic Test: measurement of multiple biomarkers

INTERVENTIONS:
Diagnostic Test: measurement of multiple biomarkers — All patients were tested for glucose and cholesterol levels. The capillary blood glucose level was measured by an electrochemical method using an Accu-Chek Active by AkkuChek blood glucose meter. The DM was considered to be verified when there were criteria which the World Health Organization (WHO) set in 2001: glucose concentration in whole blood is >6.1 mmol/l, and glucose concentration is >11.1 mmol/l in random measurement. Plasma for the study was obtained via the standard phlebotomy technique from ethylenediaminetetraacetic acid (EDTA) anticoagulants. Plasma was aliquoted into cryovials and got frozen quickly. The samples were stored in a low-temperature refrigerator (-70°C) until the study commencement (up to 3 months). All biomarkers were measured by magnetic bead-based multiplex immunofluorescence assay through the Xmap technology using the Milliplex map Human CVD Magnetic Bead Panel 1 (Millipore)

SUMMARY:
The study of biochemical risk factors for cardiovascular diseases is important not only for analysis, but also for preventive measures, given that changes in the level of biomarkers can be detected before the first clinical manifestations of CVD. Accordingly, patients at high CV risk may have additional motivation to lead a healthy lifestyle. In addition, information on biochemical risk markers can be used to optimize the clinical management of patients.

DETAILED DESCRIPTION:
Recruitment of 1500 people randomly without previous cardiovascular events. Examination, questioning of patients, laboratory tests. Patient follow-up for 6 years. Registration of the facts of the occurrence of cardiovascular events.

Cohort study with a retrospective and prospective component

Stage I (Conducted in 2014 as part of the scientific and technical project "Environmental risks and public health")

1. Questionnaire and general clinical examination (anthropometry, measurement of blood pressure, BMI, WC)
2. determination of cholesterol, glucose and total cardiovascular risk according to the SCORE scale
3. Determination of the quality of life, the level of depression and anxiety, the level of physical activity.

For an in-depth biochemical blood test for onco- and cardiomarkers, the MILLIPLEX MAP Human panel was used. This panel allows you to simultaneously study 23 onco- and 11 cardiac markers, which are the most common among oncological and cardiac diseases. Tumor markers included: alpha-fetoprotein (Afp), carbohydrate antigen 125 (CA125), carbohydrate antigen 15-3 (CA15-3), cancer embryonic antigen (CEA), cytokeratin fragment 19 (CYFRA21-1), fibroblast growth factor 2 (FGF2), human epididymis protein 4 (HE4), hepatocyte growth factor (HGF-α), interleukin 6 (IL6), interleukin 8 (IL8), leptin (LEPTIN), anti-Mullerian hormone (MIF), osteopontin (OPN ), prolactin (PROLACTIN), common prostate specific antigen (PSAtotal), cystatin C (SCF), apoptosis inducer (SFAS), transforming growth factor (TGF-α), tumor necrosis factor (TNF), TRAIL, vascular endothelial growth factor ( VEGF), Beta chorionic gonadotropin (bHCG), apoptosis inducer L (SFAS) L.

In respondents with cardiovascular risk (1% or more on the SCORE scale), the level of cardiomarkers was determined. Cardiomarkers included: creatine kinase MB (CK MB), chemokine C-X-C motif, ligand 16 (CXCL16), fatty acid binding protein, cardiac form (FABP3), N-terminal fragment of the brain natriuretic peptide (NT-ProBNP), oncostatin M (OSM), placental growth factor isoform (PIGF 4), C-X-C motif chemokine, ligand 6 (CXCL6), endocan 1 (ENDOCAN1), fatty acid binding protein 4 (FABP-4), TNF superfamily protein ( LIGHT), troponin I (TROPONINI).

Determination of the content of biochemical markers in the blood (carried out at the Collective Use Laboratory of the NJSC "Medical University of Karaganda").

STAGE II Prospective observation for 6 years, For a cardiovascular event we take the development of: Acute forms of ischemic disease (ACS with and without ST-segment elevation / myocardial infarction), chronic forms of IHD-angina pectoris, Acute cerebrovascular accident, transient ischemic attack, Lethal outcome from CVD, death from all causes.

Statistical data processing will be carried out using the SPSS program (version 22.0). Quantitative variables with a normal distribution will be presented as mean values and their standard deviations (M ± SD), with a difference from the normal distribution - median and interquartile range (Me (IQR). Dichotomous signs are presented as shares (absolute number of patients (%) Descriptive statistics will use the Mann-Whitney U-test for independent samples to compare quantitative data, categorical data will be analyzed using Pearson's χ2, Spearman's (Rho) correlation analysis will be used to determine the relationship between parameters, Using binary logistic regression (one-way and multivariate) if independent predictors of the NSS and the odds ratio (OR) are established at a 95% confidence interval (CI) for each factor.Based on the results of multivariate regression analysis on the values of exp(B) of significant variables and constants, a predictive model will be built, predictive value ( specificity, h Sensitivity, % of false positive and false negative results. Cox regression, Kaplan-Meier survival analysis will also be used, there will be a comparison of C-statistics of models. The critical level of significance (p) when testing statistical hypotheses will be taken as 0.05.

ELIGIBILITY:
iInclusion Criteria:

• respondents living in the territory of the Republic of Kazakhstan from 25 to 65 years without previous cardiovascular events.

Exclusion criteria:

* pregnant women;
* persons with mental and severe neurological diseases;
* survivors of an acute event associated with atherosclerosis;
* persons with diagnosed chronic forms of coronary artery disease;
* persons with verified CHF;
* persons with myocarditis and cardiomyopathies of various origins,
* congenital and acquired heart defects,
* atherosclerosis of peripheral arteries.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: persons living in the Republic of Kazakhstan, aged 25 to 65 years without previous cardiovascular events
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
number of respondents with stroke or transient ischemic attack | 66 months
  stroke was defined as a sudden onset of nonconvulsive and focal neurological deficit due to ischemia or hemorrhage that lasts >24 hours, and it is transient ischemic attack if neurological recovery occurred within 24 hours. &e diagnosis of stroke and the transient ischemic attack was based on the disease history, neurological examination, and all available clinical data, including computed tomography (CT)/magnetic resonance imaging (MRI) results.
Number of respondents with Coronary heart disease | 66 months
  Coronary heart disease included myocardial infarction, sudden cardiac death, and newly diagnosed angina. The criteria for MI were at least two of the following: (1) typical symptoms, including prolonged severe anterior chest pain; (2) elevated cardiac enzymes-higher than twice the upper limit of the standard values; sudden cardiac death within 1 hour of the acute condition onset; (3) progressive diagnostic electrocardiographic changes. The cases of newly diagnosed angina were determined based on typical angina-type pain, reversed by the use of nitrates, confirmed by a doctor's examination, and via the electrocardiography (ECG) exercise test.
Number Of respondents wirh cardiovascular death | 66 months
  death reported as a complication of cardiovascular disease

CONTACTS AND LOCATIONS:
Overall Officials: Lyudmila Turgunova, MD, PhD, ScD, Principal Investigator — Karaganda Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pareek M, Bhatt DL, Vaduganathan M, Biering-Sorensen T, Qamar A, Diederichsen AC, Moller JE, Hindersson P, Leosdottir M, Magnusson M, Nilsson PM, Olsen MH. Single and multiple cardiovascular biomarkers in subjects without a previous cardiovascular event. Eur J Prev Cardiol. 2017 Oct;24(15):1648-1659. doi: 10.1177/2047487317717065. Epub 2017 Jun 23. PMID 28644092
- [Result] Pauli N, Puchalowicz K, Kuligowska A, Krzystolik A, Dziedziejko V, Safranow K, Rac M, Chlubek D, Ewa Rac M. Associations between IL-6 and Echo-Parameters in Patients with Early Onset Coronary Artery Disease. Diagnostics (Basel). 2019 Nov 14;9(4):189. doi: 10.3390/diagnostics9040189. PMID 31739518
- [Result] Shi C, van der Wal HH, Sillje HHW, Dokter MM, van den Berg F, Huizinga L, Vriesema M, Post J, Anker SD, Cleland JG, Ng LL, Samani NJ, Dickstein K, Zannad F, Lang CC, van Haelst PL, Gietema JA, Metra M, Ameri P, Canepa M, van Veldhuisen DJ, Voors AA, de Boer RA. Tumour biomarkers: association with heart failure outcomes. J Intern Med. 2020 Aug;288(2):207-218. doi: 10.1111/joim.13053. Epub 2020 May 5. PMID 32372544
- [Result] Bracun V, Suthahar N, Shi C, de Wit S, Meijers WC, Klip IT, de Boer RA, Aboumsallem JP. Established Tumour Biomarkers Predict Cardiovascular Events and Mortality in the General Population. Front Cardiovasc Med. 2021 Dec 8;8:753885. doi: 10.3389/fcvm.2021.753885. eCollection 2021. PMID 34957244
- [Result] Chatzinikolaou A, Tzikas S, Lavdaniti M. Assessment of Quality of Life in Patients With Cardiovascular Disease Using the SF-36, MacNew, and EQ-5D-5L Questionnaires. Cureus. 2021 Sep 14;13(9):e17982. doi: 10.7759/cureus.17982. eCollection 2021 Sep. PMID 34667665
- [Result] Kwee LC, Neely ML, Grass E, Gregory SG, Roe MT, Ohman EM, Fox KAA, White HD, Armstrong PW, Bowsman LM, Haas JV, Duffin KL, Chan MY, Shah SH. Associations of osteopontin and NT-proBNP with circulating miRNA levels in acute coronary syndrome. Physiol Genomics. 2019 Oct 1;51(10):506-515. doi: 10.1152/physiolgenomics.00033.2019. Epub 2019 Sep 18. PMID 31530226